CLINICAL TRIAL: NCT03738046
Title: Help Overcoming Prodromal Experiences Through Early Assessment & Management - Clinical High Risk Group CBSST
Brief Title: HOPE TEAM - Clinical High Risk Group CBSST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We had a change in staffing that precluded pursing this project
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Leslie Horton, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO18010551
Record Dates: First submitted 2018-10-16; First posted 2018-11-13 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Prodromal Symptoms; Prodromal Stage; Prodromal States; Psychosis
MeSH Terms: conditions — Prodromal Symptoms; Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Treatment Arm (Experimental): Group therapy will occur once weekly (60-90-minute sessions) at the HOPE TEAM offices for 24 weeks. The group sessions with consist of 4 skill modules, each of which last 6 sessions. Three of these--the Cognitive, Social Skills, and Problem-Solving Modules-will be modules taken from Cognitive and Behavioral Social Skills Training (CBSST; Granholm McQuaid, & Holden, 2016) and modified for use with CHR adolescents. The fourth module-Stress Coping-will be adapted for this sample from an established group CBT treatment for psychosis (Lecomte, Leclerc, & Wykes, 2016).
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Group therapy will occur once weekly (60-90-minute sessions) at the HOPE TEAM offices for 24 weeks. The group sessions with consist of 4 skill modules, each of which last 6 sessions. Three of these--the Cognitive, Social Skills, and Problem-Solving Modules-will be modules taken from Cognitive and Behavioral Social Skills Training (CBSST; Granholm McQuaid, & Holden, 2016) and modified for use with CHR adolescents. The fourth module-Stress Coping-will be adapted for this sample from an established group CBT treatment for psychosis (Lecomte, Leclerc, & Wykes, 2016).
  Other Names: Cognitive Behavioral Social Skills Therapy

SUMMARY:
Community-based treatments for adolescents at risk for psychosis are not widely available, nor are there established, gold-standard psychosocial group interventions for this population. The HOPE TEAM, Helping Overcome Prodromal Experiences through Treatment and Evaluation of Adolescent Minds (PI: Bachman; funded by The Pittsburgh Foundation) is an early detection and intervention program for youth at clinical high risk for psychosis which aims to help them by engaging existing community resources, providing assessment, and offering trauma-informed psychotherapy. Embedded within the Family Care Connection Center at Turtle Creek, the HOPE TEAM offers individual psychotherapy as part of its clinical service model. The present study seeks to evaluate, in a small and preliminary sample (n = 20), the feasibility and effectiveness of a 24-week Cognitive-Behavioral Social Skills Therapy (CBSST) group intervention for CHR adolescents who are part of the HOPE TEAM. To that end, the current proposal will seek to conduct brief research assessments to assess the group members' perceptions of the group's utility, as well as their current clinical symptoms and functioning prior to, during, and after participating in this group. The goals of this pilot project are to 1) identify which aspects of the group perceived to be most and least helpful by participating adolescents, and 2) evaluate whether participation in the group meaningfully improves participants' clinical symptoms and functioning. The investigators aim to use these pilot data to guide future selection of treatment targets in this clinical practice, and to identify future strategies for increasing satisfaction and retention in community-based group interventions for CHR adolescents.

DETAILED DESCRIPTION:
Accumulating evidence suggests that psychotherapy, particularly CBT (Cognitive-Behavior Therapy) may effectively lower clinical high risk (CHR) youths' risk of developing psychosis. This is consistent with converging evidence that CBT, in both individual and group delivery formats, is effective for reducing positive symptoms of psychosis in those with a diagnosis of schizophrenia. Social Skills Training (SST) for psychosis may be more beneficial for treating negative symptoms and social impairment that accompany schizophrenia.

Given these findings, a group therapy modality combining CBT and SST (CBSST) has been developed with the goal of addressing multiple domains of symptoms and impairments; outcomes of randomized clinical trials have shown that individuals with schizophrenia who received CBSST had improved functioning and less severe psychotic symptoms.4 Furthermore, CBSST is also feasible and well accepted for adolescents and young adults with a first episode of psychosis. However, there are no established, gold-standard psychosocial group interventions for CHR youth, nor have studies specifically investigated the efficacy of CBSST for this population. Since CBSST is effective in adult psychosis, a modified version of this group treatment modality may be useful for CHR adolescents. Given the high levels of victimization, adversity, and stress in community CHR samples, modifications to CBSST for CHR youth should explicitly include a focus on stress coping.

Any clients ages 13-19 already enrolled in HOPE TEAM assessment will be informed about the availability of the HOPE Group by their individual clinician. If interested, potential participants (and their parents, if under age 18) will meet with study PI and Group Leader, to discuss the study and complete the informed consent process. As part of this process, adolescents (and their parents if under 18) will be made aware that their choice to participate or not in the HOPE Group will not affect any other services proved through the HOPE TEAM. Once a minimum of 4 participants are recruited for the HOPE group, the first session will be scheduled.

Group therapy will occur once weekly (60-90-minute sessions) at the HOPE TEAM offices for 24 weeks. The group sessions with consist of 4 skill modules, each of which last 6 sessions. Three of these--the Cognitive, Social Skills, and Problem-Solving Modules-will be modules taken from Cognitive and Behavioral Social Skills Training (CBSST) and modified for use with CHR adolescents. The fourth module-Stress Coping-will be adapted for this sample from an established group CBT treatment for psychosis.

Within 2 weeks of the first group session, participants will complete a very brief (25-40 minute) pre-group assessment battery in the HOPE Team offices with the PI, consisting of the:

* Youth Inventory 4-Self-Report (YSI-4; ages 14-17) or Adult Self-Report Inventory-4 (ASI-4; ages 18) are 128-item measures that takes approximately 10-15 minutes to complete. Assesses clinical symptoms, compared to a normed sample, across disruptive, mood, anxiety, and other clinical disorders.
* Prodromal Questionnaire, Brief Version (PQ-B); a 21- item dimensional self-report measure of psychotic symptoms, which takes approximately 5-10 minutes to complete.
* Defeatist Performance Attitudes Test, a 15-item questionnaire assessing dysfunctional attitudes commonly targeted by CBT therapy. This measure takes approximately 5 minutes to complete.
* HOPE Group Pre-Survey: A 5-item survey assessing open-ended thoughts about joining a group; takes approximately 5-10 minutes.

To allow for flexibility in the community treatment setting, the HOPE Group will adopt a modular rolling admissions approach to enrollment, in which new group members (up to a maximum group membership of 10) can be enrolled at the start of each module (every 6 sessions). In this case, the pre-group assessment battery will be completed with the participant within 2 weeks of their first group.

Each session will consist of collaborative agenda-setting, review of at-home practice, introduction of a new skill, skill practice, and assigning in-home practice/ summarizing the session. The end of each 60-90-minute group session will consist of 5 minutes of assessment. Group members will complete the:

* Modified QuickLL, a 14-item measure assessing how participants currently view themselves and their engagement in that day's group session. Each item is rated on a 3-point scale and the measure is totaled, with higher totals indicating better self-perception and greater engagement in the group. This measure takes approximately 2 minutes to complete.
* Simultaneously, both group leaders will complete the Participation Scale, a 9-item checklist assessing the participation and behavior of each group member, with each item rated from 0 (absence of behavior) to 4 (strong presence of behavior). A total score is computed for each participant, as well as an average for all group members, with higher scores indicated more group engagement and prosocial behaviors.

Within two weeks after completion of the 24-week Group, participants will complete a very brief (25-40 minute) post-group assessment battery in the HOPE Team offices with the PI, consisting of the:

* Youth Inventory 4-Self-Report, or Adult Self-Report Inventory-4
* Prodromal Questionnaire, Brief Version
* Defeatist Performance Attitudes test
* HOPE Group Post-Survey: A 5-item survey assessing open-ended thoughts about experiences in a group; takes approximately 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be included if they are 13-19 years old and receiving individual therapy or professional assessment/clinical evaluation as part of the HOPE TEAM.
* Due to the nature of the definition of "clinical high risk status," these patients may have a variety of clinical diagnoses, but all will be receiving individual therapy or clinical evaluation through the HOPE TEAM due to their elevated risk for developing a psychotic disorder.
* The individual therapy being provided to patients who are also eligible for HOPE TEAM Group may also vary based on their individual needs and therapy goals.

Exclusion Criteria:

* HOPE TEAM adolescents may be excluded if they express an unwillingness to participate in weekly group therapy and abide by group rules.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Utility of CBSST in a CHR group therapy setting | 6 months (end of group)
  The goals of this pilot project are to: 1) identify which aspects of the group perceived to be most and least helpful and relevant by participating adolescents, and 2) evaluate whether participants perceive that the group has impacted their clinical symptoms and functioning.
  To measure the perceived utility of CBSST in a CHR group therapy setting, a qualitative analysis of the open-ended HOPE Group Pre- and Post-Surveys will be conducted. In addition, the results of a Likert scale on the pre- and post- surveys will be analyzed. This scale presents examples of 7 domains of skills (e.g. "Thinking clearly") and participants are asked how much they feel the group has assisted them in improving this skill on a five-point Likert scale ("much worse" to "greatly improved").
Non-specific, CHR symptom reduction | 6 months (end of group)
  An additional goal of this pilot project is to address and reduce the number or severity of non-specific, sub-threshold symptoms of the clinical high-risk phase of psychotic disorders experienced by the group members.
  To measure symptom reduction, pre-group and post-group scores on the Youth Inventory Self-Report, or Adult-Self Report Inventory (depending on participant age) will be compared for each individual who completed group therapy. Symptom reduction is defined as a decrease in the overall total scores on the Youth Inventory Self-Report or Adult-Self Report Inventory (i.e. the number of symptoms reported by participants).

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Horton, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No